CLINICAL TRIAL: NCT00736216
Title: Knowledge and Perceptions About Human Papillomavirus and Cervical Cancer Risk Among Young Adults
Status: Withdrawn | Type: Observational
Why Stopped: PI left the institution
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE11806; P30CA043703 (NIH); CASE11806 (Other: Case Comprehensive Cancer Center); CASE-11806-CC231
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; human papilloma virus infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: survey administration — Participants complete the Young Adult Survey online documenting demographic data; sexual history (i.e., whether they ever had sex, age of first sexual encounter, number of life time partners, condom use, sexually transmitted diseases [STDs], and pregnancy history); cigarette use; current and past drug use; knowledge of human papillomavirus (HPV) and cervical cancer; past history of Pap tests and STD screenings; attitudes towards HPV testing; vaccine knowledge and acceptability; sources of information about HPV; source of information about cervical cancer; identification of common STDs; perceived risk of acquiring STDs; perceived risk of acquiring HPV; social support; and religion.

SUMMARY:
RATIONALE: Learning about young adults' knowledge and perceptions about risk factors for the human papilloma virus and cervical cancer may help doctors learn more about how to prevent human papilloma virus infection and cervical cancer in the future.

PURPOSE: This clinical trial is studying knowledge and perceptions of the risk factors for human papilloma virus infection and cervical cancer in young adults.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the socio-demographic context of college students in an urban Midwestern setting.
* Assess knowledge of the human papillomavirus (HPV) and cervical cancer in these participants.
* Assess the population's perception of HPV risk.
* Assess the prevalence of risk behaviors that may place this population at risk for HPV.
* Identify the best predictors of HPV knowledge and cervical cancer knowledge.
* Assess vaccine knowledge and acceptance in these participants.

OUTLINE: Participants complete the Young Adult Survey online documenting demographic data; sexual history (i.e., whether they ever had sex, age of first sexual encounter, number of life time partners, condom use, sexually transmitted diseases [STDs], and pregnancy history); cigarette use; current and past drug use; knowledge of human papillomavirus (HPV) and cervical cancer; past history of Pap tests and STD screenings; attitudes towards HPV testing; vaccine knowledge and acceptability; sources of information about HPV; source of information about cervical cancer; identification of common STDs; perceived risk of acquiring STDs; perceived risk of acquiring HPV; social support; and religion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently enrolled in a college, university, or community college in the Greater Cleveland metropolitan area
* Currently single and never married

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community based outreach in an urban Mid-west area
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Socio-demographic context of college students in an urban Midwestern setting
Knowledge of human papillomavirus (HPV) and cervical cancer
Perception of HPV risk
Prevalence of risk behaviors that may place this population at risk for HPV
Best predictors of HPV knowledge and cervical cancer knowledge
Vaccine knowledge and acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A. Francis, PhD, MPH, CHES, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (8):
- United States (8):
  - Geauga Regional Hospital, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Cleveland, Ohio